CLINICAL TRIAL: NCT07328919
Title: A Phase III, Randomized Controlled, Open-Label, Multicenter Clinical Study Evaluating the Efficacy and Safety of TT-00420 Tablets Versus Chemotherapy in Patients With Surgically Unresectable Advanced or Metastatic Intrahepatic Cholangiocarcinoma Harboring FGFR2 Fusions/Rearrangements or Mutations, Who Have Progressed or Relapsed After Prior First-Line Systemic Therapy
Brief Title: Efficacy and Safety of TT-00420 (Tinengotinib) Tablets Versus Chemotherapy in Patients With Advanced Intrahepatic Cholangiocarcinoma Harboring FGFR2 Fusions/Rearrangements or Mutations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT00420CN18
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Advanced Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (TT-00420 monotherapy) (Experimental): The starting dose of TT-00420 tablets is 10 mg QD (5 mg per tablet, 2 tablets), administered orally and taken continuously.
  Interventions: Drug: TT-00420 (tinengotinib)
- Arm B (chemotherapy) (Active Comparator): Chemotherapy includes mFOLFOX regimen, XELIRI regimen or irinotecan monotherapy.
  Interventions: Drug: Oxaliplatin, fluorouracil, calcium folinate, irinotecan, capecitabine

INTERVENTIONS:
Drug: TT-00420 (tinengotinib) — Subject will receive TT-00420 (tinengotinib) once daily in 28-day cycles with initial dosage of 10 mg QD per protocol defined schedule.
  Arms: Arm A (TT-00420 monotherapy)
Drug: Oxaliplatin, fluorouracil, calcium folinate, irinotecan, capecitabine — Subjects will receive chemotherapy (mFOLFOX regimen, XELIRI regimen, or irinotecan monotherapy). The dosing schedule involves intravenous administration or oral intake every two weeks (except for capecitabine). Treatment continues until the occurrence of confirmed disease progression, intolerable toxicities, withdrawal of informed consent, death, or other reasons specified in the protocol (whichever occurs first). Among these, subjects receiving the mFOLFOX regimen are limited to a maximum of 6 treatment cycles (approximately 12 administrations).
  Arms: Arm B (chemotherapy)

SUMMARY:
This is an open-label, randomized, controlled, multicenter, phase III clinical study designed to evaluate the efficacy and safety of TT-00420 tablets as monotherapy versus chemotherapy in subjects with unresectable advanced or metastatic intrahepatic cholangiocarcinoma harboring FGFR2 gene fusions/rearrangements or mutations, who have experienced recurrence or progression after prior first-line systemic chemotherapy.

DETAILED DESCRIPTION:
Approximately 138 subjects will be enrolled. Eligible subjects will be randomized in a 2:1 ratio to one of the two arms: Arm A (TT-00420 tablet monotherapy) or Arm B (chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed intrahepatic cholangiocarcinoma.
3. Subjects diagnosed with stage III or IV intrahepatic cholangiocarcinoma according to the American Joint Committee on Cancer (AJCC) 8th Edition (2018) staging system, and assessed by the investigator as not eligible for curative surgical resection.
4. Subjects who have experienced recurrence or progression after receiving only one prior line of systemic chemotherapy combined with immunotherapy (PD-1/PD-L1 inhibitor), with or without targeted therapy. Sequential immunotherapy following the completion of chemotherapy cycles is also considered part of the first-line combined regimen. First-line systemic chemotherapy is defined as gemcitabine/capecitabine with or without a platinum-based agent.

   Note: Recurrence within 6 months after completion of adjuvant or neoadjuvant therapy will be considered as a line of systemic therapy. Local treatments do not count as systemic therapy.
5. The presence of FGFR2 gene fusion/rearrangement or mutation must be confirmed by detection using tumor tissue samples provided by the patient and analyzed by a central laboratory.
6. At least one radiographically measurable lesion must be present according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. ECOG ≤ 1.
8. Subjects must have adequate organ and bone marrow function.

Exclusion Criteria:

1. Subjects with a history of prior treatment with TT-00420 tablets.
2. Subjects with a known severe allergic reaction to any agent in the study and for whom no alternative study treatment is available.
3. Subjects receiving corticosteroid therapy for CNS metastases are also ineligible.
4. Concurrent active malignancy requiring active treatment. Malignancies diagnosed >5 years ago without the need for treatment, as well as cured localized tumors such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, or papillary thyroid carcinoma, are allowed.
5. Administration of other anti-tumor drugs prior to randomization with an interval of ≤ 5 half-lives or 14 days (whichever is shorter), or failure to recover from adverse events of prior therapies (except for adverse events of ≤ Grade 1, or ≤ Grade 2 events judged by the investigator as not constituting a safety risk).
6. Prior radiation therapy (large-field radiotherapy within 4 weeks, or local palliative radiotherapy within 2 weeks, before randomization), or failure to recover from related adverse events, is excluded. However, initiation of the investigational drug during the washout period is permitted with sponsor approval, if the investigator believes it is in the subject's best interest based on a favorable benefit-risk assessment.
7. Subjects who have undergone major surgery within 4 weeks prior to randomization, or who have not recovered from related adverse events (with the exception of ≤ Grade 1 events or non-risk Grade 2 events per investigator's judgment), are excluded.
8. Subjects with uncontrolled hypertension (defined as blood pressure of ≥ 150 mm Hg systolic and/or ≥ 90 mm Hg diastolic despite adequate treatment with antihypertensive medications at screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS by BICR | From first study drug administration until the date of first documented progression assessed by BICR or date of death from any cause, whichever came first, assessed up to 24 months.
  Progression-free survival (PFS) by BICR: PFS is defined as the time from date of randomization to the date of first documented disease progression as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or date of death due to any cause, whichever is earlier.

SECONDARY OUTCOMES:
Overall Survival (OS) | From first study drug administration until the date of death from any cause, assessed up to 24 months.
  OS is defined as the time from date of randomization to date of death of any cause.
PFS by Investigators per RECIST v1.1. | From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  PFS is defined as the time from date of randomization to the date of first documented disease progression as assessed by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Objective Response Rate (ORR) by BICR and by Investigator | Through study completion, an average of 9 months.
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Duration of Response (DOR) by BICR and by Investigator | Through study completion, an average of 9 months.
  Duration of response for CR or PR based on RECIST version 1.1.
Disease Control Rate (DCR) | Through study completion, an average of 9 months.
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) or a stable disease (SD) based on RECIST version 1.1.
Incidence, duration, and severity of adverse events (AEs) | Up to 30 days from study discontinuation.
  As assessed per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (or the most current version).

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Eastern Hepatobiliary Surgery Hospital, Shanghai
  - Fudan University Shanghai Cancer Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No